CLINICAL TRIAL: NCT06705816
Title: Cognitive Function in Rett Syndrome During Trofinetide Treatment
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 33488
Record Dates: First submitted 2024-11-11; First posted 2024-11-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with Rett Syndrome who are interested in Trofinetide treatment
  Interventions: Other: None interventional

INTERVENTIONS:
Other: None interventional — This is an observational study

SUMMARY:
Assessing cognitive functions among individuals with severe intellectual and developmental disabilities (IDD), including RTT, is often challenging due to floor effects of many standardized assessment batteries in this population. In addition, deficits in motor function and verbal ability may obscure certain abilities in this population when using standard IQ measures. Remote eye-tracking tasks have been proposed as an alternative approach for assessing cognitive functions among individuals with severe IDD, because eye-tracking tasks can be designed to minimize the influence of gross motor and receptive language deficits on performance. Although several types of eye-tracking tasks have been evaluated in RTT, most have been implemented only at a single time-point. As a result, it is unclear whether these measures are stable over time, or sensitive to developmental changes or alterations to health status that occur in RTT (e.g., developmental regression, development of seizures, change in medication, etc.). With the recent FDA approval of trofinetide for the treatment of RTT, we have a novel opportunity to test the sensitivity of eye-tracking and other psychophysiological measures to treatment changes. Anecdotally, parents and clinicians have reported improvements in attention and alertness during trofinetide treatment, but currently available outcome measures do not capture these types of effects. Therefore, we propose to conduct a pilot trial of changes in measures of attention, oculomotor function, learning, and autonomic function, all collected using non-invasive measures, during trofinetide treatment. This is an observational within-subject design with a 4-week post-treatment assessment compared to two pre-treatment assessments. Additional optional follow-up assessments will be performed with families who are interested and returning for standard-of-care visits to Gillette or who are willing to travel for a research-only visit.

ELIGIBILITY:
Inclusion Criteria:

* Any individuals who are initiating trofinetide treatment for RTT through the physicians associated with the Gillette Children's RTT clinic will be potentially eligible for participation, regardless of age. To enroll, participants must meet the following criteria:

  1. Provision of signed and dated informed consent form by the individual's parent/legal guardian
  2. Stated willingness to comply with all study procedures and availability for the duration of the study
  3. Documented diagnosis of Rett syndrome
  4. Participant is not showing active signs of developmental regression, defined as: no loss or degradation of ambulation within the past 6 months; no loss or degradation of hand function within the past 6 months; and no loss or degradation of verbal or non-verbal communication or social skills in the past 6 months.
  5. Participant's current pharmacological treatment regimen has been stable for at least 4 weeks.
  6. Seeking prescription for trofinetide through the Gillette Children's Rett syndrome clinic

Exclusion Criteria:

1. Diagnosis of a progressive medical or neurological condition that in the opinion of the investigator would interfere with the conduct of the study.
2. Current clinically significant systemic illness that is likely to result in the deterioration of the participant's condition during the study.
3. Participants taking any other investigational drug currently or within the past 30 days.
4. Known, uncorrected visual impairment that would limit the ability to view images during eye-tracking tasks.
5. Severe behavioral problems (i.e., aggression, property destruction, extreme hyperactivity) that would interfere with participation in study activities.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any individuals who are initiating trofinetide treatment for RTT through the physicians associated with the Gillette Children's RTT clinic will be potentially eligible for participation, regardless of age.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function in Rett Syndrome During Trofinetide Treatment | baseline, 6weeks to 12 months
  change in saccade latencies during the 'statistical learning' paradigm
Eye movement gaze fixations | baseline, 6weeks to 12 months
  change in duration of gaze fixation to the correct image during the 'Looking While Listening' paradigm.

SECONDARY OUTCOMES:
Heart rate variability | baseline, 6weeks to 12 months
  Change in baseline heart rate variability during sustained attention during eye-tracking tasks.
Heart rate suppression | baseline, 6weeks to 12 months
  Change in baseline heart rate suppression during sustained attention during eye-tracking tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States